CLINICAL TRIAL: NCT05486533
Title: The Effect of Acupressure After Angiography on Pain Level and Hemodynamic Variables Randomized Controlled Study
Brief Title: The Effect of Acupressure After Angiography on Pain Level and Hemodynamic Variables
Acronym: Acupress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Tugba CAM YANIK, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersinUnive
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Acupressure; Pain; Hemodynamic Instability; Angiopathy, Peripheral
MeSH Terms: conditions — Pain; Peripheral Vascular Diseases | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, three-arm randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the research, participants and researchers cannot be blinded. Analyzes will be made by a biostatistician independent of the research and the statistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will be given acupressure.
  Interventions: Other: Acupressure
- Control (No Intervention): It will only take routine treatment and care.

INTERVENTIONS:
Other: Acupressure — The experimental group will start with LI4 points and continue P6 and LI11 points. The application will be carried out by determining the priority order of the points with the draw. Attention will be paid to the intensity and duration of the pressure deemed appropriate. Since the individuals' responses will differ, the stiffness and pressure will be adjusted according to the individual's sensitivity not to cause tissue damage. Before starting the application, around the area to be pressed for 20-30 seconds will be gently rubbed with palm. With the gentle rubbing of the surrounding tissue, the tension and tissue sensitivity in warming, relaxing and preparatory will be reduced, and the tissue will be relieved. After, the point determined will be pressed manually for 2 minutes.
  Other Names: Acupress
  Arms: Experimental

SUMMARY:
This randomized controlled study evaluates the effect of acupressure application on the pain level patients after angioography. The hypothesis of this study is that acupressure reduces pain levels and stabilizes hemodynamic variables.

DETAILED DESCRIPTION:
In the study, 124 patients will randomly assigned to acupressure/experimental group and control group. To the acupressure/experimental group (n = 62), an average of 15 minutes will be applied to the LI4 (liver, between thumb and forefinger), P6 (pericardium, three fingers above the wrist) and LI 11 is located the area where the elbow bend. On the other hand, no other intervention will be applied to the control group other than routine treatment and nursing care. The primary outcome of the research is the effect of acupressure on the pain of patients. The secondary outcome of the study is to determine the effect of acupressure on the hemodynamic variables. The pain and hemodynamic variables will be collected before, immediately after the application, 10th, 20th and 30th minutes after the application. Data will also be collected from the control group at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research (signing the Informed Consent Form),
* Conscious and cooperative,
* Speaks and understands Turkish,
* Over 18 years of age,
* Stable general condition,
* No sensitivity in the area where acupressure will be applied,
* No active COVID-19 infection,
* Patients without any psychiatric diagnosis will be included.

Exclusion Criteria:

* Do not agreeing to participate in the research (signing the Informed Consent Form),
* Do not conscious and cooperative,
* Do not speaks and understands Turkish,
* Do not over 18 years of age,
* Do not stable general condition,
* Having sensitivity in the area where acupressure will be applied,
* Having active COVID-19 infection,
* Patients with any psychiatric diagnosis will be included.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Pain evaluated using the visual analog scale | Change from before implementation and immediately after, 10th, 20th and 30th minutes after implementation
  The total scale score is in the range of 0 cm (minimum) -10 cm (maximum). A score of 0 indicates no pain and a score of 10 indicates very severe pain.

SECONDARY OUTCOMES:
Systolic blood pressure | Change from before implementation and immediately after, 10th, 20th and 30th minutes after implementation
  Systolic blood pressure (SBP), mmHg
Diastolic blood pressure | Change from before implementation and immediately after, 10th, 20th and 30th minutes after implementation
  Diastolic blood pressure (DBP), mmHg
Heart rate | Change from before implementation and immediately after, 10th, 20th and 30th minutes after implementation
  Beats per minute
Respiratory rate | Change from before implementation and immediately after, 10th, 20th and 30th minutes after implementation
  Lung breathing
Peripheral oxygen saturation | Change from before implementation and immediately after, 10th, 20th and 30th minutes after implementation
  %, percentage of oxygenated hemoglobin in peripheral arterial blood

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Altun Uğraş, PhD, Study Director — Mersin University; Canan KANAT, Master, Principal Investigator — Mersin University; Barış DÜZEL, Specialist, Principal Investigator — Mersin City Research and Application Hospital
Locations (1):
- Turkey, Mersin University,, Mersin, Turkey/Mersin,Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajaee, N., Choopani, N., Pishgoei, A. H., & Sharififar, S. (2015). The effect of acupressure on Patient's anxiety who candidate for coronary angiography. Military Caring Sciences, 1 (3), 6-13.
- [Result] The effect of acupressure on vital signs, acute pain, stress and satisfaction during venipuncture: Single-blind, randomized controlled study. European